CLINICAL TRIAL: NCT01021852
Title: A Phase IIb, Multicenter, Randomized, Double-Blind, Placebo-Controlled, 2-Period Adaptive Crossover Polysomnography Study to Evaluate the Safety and Efficacy of MK-6096 in Patients With Primary Insomnia
Brief Title: Polysomnography Study of MK-6096 in Participants With Primary Insomnia (MK-6096-011)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 6096-011; MK-6096-011 (Other: Merck Registration Number)
Record Dates: First submitted 2009-11-25; First posted 2009-11-30 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-10

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — MK-6096

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- MK-6096 2.5 mg/Placebo (Experimental): Prior to Treatment Period 1, participants undergo a 3 week screening period and receive single-blind placebo for the last 2 weeks if screening criteria are met. During Treatment Period 1, participants receive MK-6096 2.5 mg daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory on Days 1 and 29 for overnight polysomnography (PSG) recordings, on which days they receive MK-6096 30 minutes before bedtime. Treatment Period 1 is followed by a 2-week washout period during which the participant receives single-blind placebo for the first 3 days and no treatment for the remaining 11 days. During Treatment Period 2, participants receive dose-matched placebo to MK-6096 daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory for 2 overnight PSG recordings on Days 1 and 29 (Study Days 44 and 72), on which days they receive placebo 30 minutes before bedtime.
  Interventions: Drug: MK-6096; Drug: Dose-matched Placebo to MK-6096
- Placebo/MK-6096 2.5 mg (Experimental): Prior to Treatment Period 1, participants undergo a 3 week screening period and receive single-blind placebo for the last 2 weeks if screening criteria are met. During Treatment Period 1, participants receive matched placebo to MK-6096 daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory for 2 overnight PSG recordings on Days 1 and 29, on which days they receive placebo 30 minutes before bedtime. Treatment Period 1 is followed by a 2-week washout period during which the participant receives single-blind placebo for the first 3 days and no treatment for the remaining 11 days. During Treatment Period 2, participants receive MK-6096 2.5 mg daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory for 2 overnight PSG recordings on Days 1 and 29 (Study Days 44 and 72), on which days they receive MK-6096 30 minutes before bedtime.
  Interventions: Drug: MK-6096; Drug: Dose-matched Placebo to MK-6096
- MK-6096 5 mg/Placebo (Experimental): Prior to Treatment Period 1, participants undergo a 3 week screening period and receive single-blind placebo for the last 2 weeks if screening criteria are met. During Treatment Period 1, participants receive MK-6096 5 mg daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory on Days 1 and 29 for 2 overnight PSG recordings, on which days they receive MK-6096 30 minutes before bedtime. Treatment Period 1 is followed by a 2-week washout period during which the participant receives single-blind placebo to MK-6096 for the first 3 days and no treatment the remaining 11 days. During Treatment Period 2, participants receive matched placebo to MK-6096 daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory for 2 overnight PSG recordings on Days 1 and 29 (Study Days 44 and 72), on which days they receive placebo 30 minutes before bedtime.
  Interventions: Drug: MK-6096; Drug: Dose-matched Placebo to MK-6096
- Placebo/MK-6096 5 mg (Experimental): Prior to Treatment Period 1, participants undergo a 3 week screening period and receive single-blind placebo for the last 2 weeks if screening criteria are met. During Treatment Period 1, participants receive matched placebo to MK-6096 daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory for 2 overnight PSG recordings on Days 1 and 29, on which days they receive placebo 30 minutes before bedtime. Treatment Period 1 is followed by a 2-week washout period during which the participant receives single-blind placebo for the first 3 days and no treatment the remaining 11 days. During Treatment Period 2, participants receive MK-6096 5 mg daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory for 2 overnight PSG recordings on Days 1 and 29 (Study Days 44 and 72), on which days they receive MK-6096 30 minutes before bedtime.
  Interventions: Drug: MK-6096; Drug: Dose-matched Placebo to MK-6096
- MK-6096 10 mg/Placebo (Experimental): Prior to Treatment Period 1, participants undergo a 3 week screening period and receive single-blind placebo for the last 2 weeks if screening criteria are met. During Treatment Period 1, participants receive MK-6096 10 mg daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory on Days 1 and 29 for 2 overnight PSG recordings, on which days they receive MK-6096 30 minutes before bedtime. Treatment Period 1 is followed by a 2-week washout period during which the participant receives single-blind placebo to MK-6096 for the first 3 days and no treatment the remaining 11 days. During Treatment Period 2, participants receive matched placebo to MK-6096 daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory for 2 overnight PSG recordings on Days 1 and 29 (Study Days 44 and 72), on which days they receive placebo 30 minutes before bedtime.
  Interventions: Drug: MK-6096; Drug: Dose-matched Placebo to MK-6096
- Placebo/MK-6096 10 mg (Experimental): Prior to Treatment Period 1, participants undergo a 3 week screening period and receive single-blind placebo for the last 2 weeks if screening criteria are met. During Treatment Period 1, participants receive matched placebo to MK-6096 daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory for 2 overnight PSG recordings on Days 1 and 29, on which days they receive placebo 30 minutes before bedtime. Treatment Period 1 is followed by a 2-week washout period during which the participant receives single-blind placebo for the first 3 days and no treatment the remaining 11 days. During Treatment Period 2, participants receive MK-6096 10 mg daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory for 2 overnight PSG recordings on Days 1 and 29 (Study Days 44 and 72), on which days they receive MK-6096 30 minutes before bedtime.
  Interventions: Drug: MK-6096; Drug: Dose-matched Placebo to MK-6096
- MK-6096 20 mg/Placebo (Experimental): Prior to Treatment Period 1, participants undergo a 3 week screening period and receive single-blind placebo for the last 2 weeks if screening criteria are met. During Treatment Period 1, participants receive MK-6096 20 mg daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory on Days 1 and 29 for 2 overnight PSG recordings, on which days they receive MK-6096 30 minutes before bedtime. Treatment Period 1 is followed by a 2-week washout period during which the participant receives single-blind placebo to MK-6096 for the first 3 days and no treatment the remaining 11 days. During Treatment Period 2, participants receive matched placebo to MK-6096 daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory for 2 overnight PSG recordings on Days 1 and 29 (Study Days 44 and 72), on which days they receive placebo 30 minutes before bedtime.
  Interventions: Drug: MK-6096; Drug: Dose-matched Placebo to MK-6096
- Placebo/MK-6096 20 mg (Experimental): Prior to Treatment Period 1, participants undergo a 3 week screening period and receive single-blind placebo for the last 2 weeks if screening criteria are met. During Treatment Period 1, participants receive matched placebo to MK-6096 daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory for 2 overnight PSG recordings on Days 1 and 29, on which days they receive placebo 30 minutes before bedtime. Treatment Period 1 is followed by a 2-week washout period during which the participant receives single-blind placebo for the first 3 days and no treatment the remaining 11 days. During Treatment Period 2, participants receive MK-6096 20 mg daily for 4 weeks at 5-10 minutes before bedtime and return to the sleep laboratory for 2 overnight PSG recordings on Days 1 and 29 (Study Days 44 and 72), on which days they receive MK-6096 30 minutes before bedtime.
  Interventions: Drug: MK-6096; Drug: Dose-matched Placebo to MK-6096

INTERVENTIONS:
Drug: MK-6096 — MK-6096 2.5 mg or 5 mg tablets equaling 2.5 mg dose, 5 mg dose, 10 mg dose, or 20 mg dose (depending upon allocation) were taken daily before bedtime for 4 weeks.
Drug: Dose-matched Placebo to MK-6096 — Dose-matched placebo tablets to MK-6096 were taken daily before bedtime during 2-week single-blind run-in, for 4 weeks as a treatment period, and during 2-week washout between treatment periods.

SUMMARY:
This was a cross-over, polysomnography (PSG) study to test the safety, tolerability and effectiveness of different doses of MK-6096 in the treatment of participants with primary insomnia. The primary efficacy hypothesis was that at least one dose of MK-6096 is superior to placebo in improving sleep efficiency (SE) as measured by PSG on Night 1 and at the end of 4 weeks of treatment (Week 4).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing to stay overnight at a sleep laboratory on 6 separate nights and is willing to stay in bed for at least 8 hours each night while at the sleep laboratory
* Participant's regular bedtime is between 9 PM and 12 AM (midnight)
* Participant is able to read and complete questionnaires and diaries
* Participant is willing to refrain from napping during the study

Exclusion Criteria:

* If female, participant is breast feeding, pregnant, or planning to become pregnant
* Participant is expecting to donate eggs or sperm during the study
* Participant has any history of a neurological disorder
* Participant has a history within the past 6 months of a cardiovascular disorder such as unstable angina, congestive heart failure or acute coronary syndrome.
* Participant has difficulty sleeping due to a medical condition
* Participant has donated blood products within the 8 weeks prior to the study
* Participant plans to travel across 3 or more time zones during the study
* Participant is currently participating or has participated in a study with an investigational compound or device within the last 30 days

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 326 (Actual)
Dates: Start 2009-11-30 (Actual); Primary Completion 2011-02-01 (Actual); Study Completion 2011-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Connor KM, Mahoney E, Jackson S, Hutzelmann J, Zhao X, Jia N, Snyder E, Snavely D, Michelson D, Roth T, Herring WJ. A Phase II Dose-Ranging Study Evaluating the Efficacy and Safety of the Orexin Receptor Antagonist Filorexant (MK-6096) in Patients with Primary Insomnia. Int J Neuropsychopharmacol. 2016 Aug 12;19(8):pyw022. doi: 10.1093/ijnp/pyw022. Print 2016 Aug. PMID 26979830
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=6096-011&kw=6096-011&tab=access

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 326 participants were randomized in this study into one of 8 treatment sequences. Participants received double-blind study drug in Treatment Period (TP)1, followed by a washout period (3 day single-blind placebo plus 11 day drug holiday), and then double-blind study drug in TP2.
Period: Treatment Period 1
Arm/Group | MK-6096 2.5 mg/Placebo | Placebo/MK-6096 2.5 mg | MK-6096 5 mg/Placebo | Placebo/MK-6096 5 mg | MK-6096 10 mg/Placebo | Placebo/MK-6096 10 mg | MK-6096 20 mg/Placebo | Placebo/MK-6096 20 mg
Started | 40 | 40 | 41 | 40 | 42 | 41 | 41 | 41
Treated | 40 | 40 | 41 | 38 | 42 | 41 (1 participant discontinued Treatment Period 1 (AE) but continued in Placebo Washout) | 41 | 41
Completed | 37 | 39 | 39 | 38 | 39 | 39 | 41 | 40
Not Completed | 3 | 1 | 2 | 2 | 3 | 2 | 0 | 1
Not completed — Adverse Event | 3 | 1 | 1 | 0 | 2 | 2 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Not Treated | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Period: Washout Period-Placebo
Arm/Group | MK-6096 2.5 mg/Placebo | Placebo/MK-6096 2.5 mg | MK-6096 5 mg/Placebo | Placebo/MK-6096 5 mg | MK-6096 10 mg/Placebo | Placebo/MK-6096 10 mg | MK-6096 20 mg/Placebo | Placebo/MK-6096 20 mg
Started | 37 | 39 | 39 | 38 | 40 (Includes 1 participant that discontinued Treatment Period 1 (AE).) | 39 (Excludes 1 participant who completed Treatment Period 1 but missed Placebo Washout) | 41 | 40
Completed | 37 | 39 | 39 | 37 | 39 | 38 | 40 | 40
Not Completed | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Washout Period-No Drug
Arm/Group | MK-6096 2.5 mg/Placebo | Placebo/MK-6096 2.5 mg | MK-6096 5 mg/Placebo | Placebo/MK-6096 5 mg | MK-6096 10 mg/Placebo | Placebo/MK-6096 10 mg | MK-6096 20 mg/Placebo | Placebo/MK-6096 20 mg
Started | 38 (Includes 1 participant who discontinued Treatment Period 1 (AE) and missed Placebo Washout.) | 39 | 39 | 37 | 39 | 39 (Includes 1 participant who completed Treatment Period 1 but missed Placebo Washout.) | 40 | 40
Completed | 37 | 39 | 39 | 37 | 39 | 38 | 40 | 40
Not Completed | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Treatment Period 2
Arm/Group | MK-6096 2.5 mg/Placebo | Placebo/MK-6096 2.5 mg | MK-6096 5 mg/Placebo | Placebo/MK-6096 5 mg | MK-6096 10 mg/Placebo | Placebo/MK-6096 10 mg | MK-6096 20 mg/Placebo | Placebo/MK-6096 20 mg
Started | 37 | 39 | 39 | 37 | 39 | 38 | 40 | 40
Completed | 37 | 38 | 38 | 37 | 37 | 37 | 37 | 38
Not Completed | 0 | 1 | 1 | 0 | 2 | 1 | 3 | 2
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-6096 2.5 mg/Placebo | Placebo/MK-6096 2.5 mg | MK-6096 5 mg/Placebo | Placebo/MK-6096 5 mg | MK-6096 10 mg/Placebo | Placebo/MK-6096 10 mg | MK-6096 20 mg/Placebo | Placebo/MK-6096 20 mg | Total
Number analyzed (Participants) | 40 | 40 | 41 | 40 | 42 | 41 | 41 | 41 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (11.9) | 47.9 (11.7) | 44.7 (10.7) | 47.6 (10.4) | 45.4 (9.9) | 45.2 (11.0) | 49.8 (9.8) | 47.0 (12.3) | 46.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 26 | 25 | 26 | 26 | 25 | 25 | 203
  Male | 15 | 15 | 15 | 15 | 16 | 15 | 16 | 16 | 123

OUTCOME MEASURES:

1. Primary Outcome: Sleep Efficiency (SE) on Night 1 and After 4 Weeks of Treatment
Description: SE was measured using a polysomnogram (PSG), which consisted of an electroencephalogram (EEG) for registration of brain activity during sleep, an electro-oculogram (EOG) for registration of the eye movements during sleep, and an electromyogram (EMG) for recording chin muscle activity during sleep. Sleep stage scoring was performed visually in 30-second epochs according to Rechtschaffen and Kales (R&K) criteria and PSG data were read by a Central Reader. SE was defined as total sleep time (TST) in minutes divided by time in bed (measured from lights off to lights on; fixed at 8 hours on each PSG night) in minutes, multiplied by 100, where TST is defined as the total time (minutes) in Stages 1, 2, 3, 4 and Rapid Eye Movement (REM). SE= (total sleep time/time in bed) x 100. Least squares (LS) mean SE was reported for each treatment arm.
Time Frame: Night 1 and end of Week 4
Population: Full Analysis Set (FAS) population; subset of all randomized participants who received at least one dose of study medication and had any post-randomization SE efficacy assessment data. The FAS population may have varied across endpoints due to the degree of missing data for each endpoint.
Measure: Least Squares Mean (Standard Error); unit: percentage of time in bed spent sleeping
Groups:
- Placebo: Participants received dose-matched placebo to MK-6096 prior to bedtime for 4 weeks (Days 1-29) during a treatment period. Placebo data were pooled across the four 2-period cross-overs within the study.
- MK-6096 2.5 mg: Participants received MK-6096 2.5 mg prior to bedtime for 4 weeks (Days 1-29) during a treatment period.
- MK-6096 5 mg: Participants received MK-6096 5 mg prior to bedtime for 4 weeks (Days 1-29) during a treatment period.
- MK-6096 10 mg: Participants received MK-6096 10 mg prior to bedtime for 4 weeks (Days 1-29) during a treatment period.
- MK-6096 20 mg: Participants received MK-6096 20 mg prior to bedtime for 4 weeks (Days 1-29) during a treatment period.
Arm/Group | Placebo | MK-6096 2.5 mg | MK-6096 5 mg | MK-6096 10 mg | MK-6096 20 mg
Number analyzed (Participants) | 313 | 79 | 78 | 80 | 80
percentage of time in bed spent sleeping
  Night 1 (n=313, 79, 78, 80, 80) | 74.8 (0.71) | 83.3 (1.54) | 84.8 (1.55) | 85.6 (1.53) | 88.2 (1.53)
  Week 4 (n=300, 76, 76, 76, 75) | 77.0 (0.71) | 81.6 (1.42) | 81.1 (1.42) | 86.7 (1.43) | 85.7 (1.43)
Statistical Analysis 1: Comparison: Placebo vs MK-6096 2.5 mg; MK-6096 2.5 mg vs. Placebo at Night 1 A mixed effects model with terms for baseline value, geographic region (Japan vs. ex-Japan), gender, treatment, sequence, period, time, and treatment-by-time interaction and period-by-time interaction was used to estimate LS mean differences between MK-6096 and placebo at Night 1. 95% confidence interval estimate and p-value (based upon a normal approximation) were also computed from the LS mean differences and variability estimates from the model; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = 8.4, 95% CI 2-sided [5.3 to 11.5], Standard Error of Mean 1.59
Statistical Analysis 2: Comparison: Placebo vs MK-6096 5 mg; MK-6096 5 mg vs. Placebo at Night 1 A mixed effects model with terms for baseline value, geographic region (Japan vs. ex-Japan), gender, treatment, sequence, period, time, and treatment-by-time interaction and period-by-time interaction was used to estimate LS mean differences between MK-6096 and placebo at Night 1. 95% confidence interval estimate and p-value (based upon a normal approximation) were also computed from the LS mean differences and variability estimates from the model; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = 9.9, 95% CI 2-sided [6.8 to 13.1], Standard Error of Mean 1.59
Statistical Analysis 3: Comparison: Placebo vs MK-6096 10 mg; MK-6096 10 mg vs. Placebo at Night 1 A mixed effects model with terms for baseline value, geographic region (Japan vs. ex-Japan), gender, treatment, sequence, period, time, and treatment-by-time interaction and period-by-time interaction was used to estimate LS mean differences between MK-6096 and placebo at Night 1. 95% confidence interval estimate and p-value (based upon a normal approximation) were also computed from the LS mean differences and variability estimates from the model; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = 10.7, 95% CI 2-sided [7.7 to 13.8], Standard Error of Mean 1.57
Statistical Analysis 4: Comparison: Placebo vs MK-6096 20 mg; MK-6096 20 mg vs. Placebo at Night 1 A mixed effects model with terms for baseline value, geographic region (Japan vs. ex-Japan), gender, treatment, sequence, period, time, and treatment-by-time interaction and period-by-time interaction was used to estimate LS mean differences between MK-6096 and placebo at Night 1. 95% confidence interval estimate and p-value (based upon a normal approximation) were also computed from the LS mean differences and variability estimates from the model; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = 13.4, 95% CI 2-sided [10.3 to 16.5], Standard Error of Mean 1.57
Statistical Analysis 5: Comparison: Placebo vs MK-6096 2.5 mg; MK-6096 2.5 mg vs. Placebo at Week 4 A mixed effects model with terms for baseline value, geographic region (Japan vs. ex-Japan), gender, treatment, sequence, period, time, and treatment-by-time interaction and period-by-time interaction was used to estimate LS mean differences between MK-6096 and placebo at Week 4. 95% confidence interval estimate and p-value (based upon a normal approximation) were also computed from the LS mean differences and variability estimates from the model; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; Difference in LS Means = 4.6, 95% CI 2-sided [1.8 to 7.4], Standard Error of Mean 1.42
Statistical Analysis 6: Comparison: Placebo vs MK-6096 5 mg; MK-6096 5 mg vs. Placebo at Week 4 A mixed effects model with terms for baseline value, geographic region (Japan vs. ex-Japan), gender, treatment, sequence, period, time, and treatment-by-time interaction and period-by-time interaction was used to estimate LS mean differences between MK-6096 and placebo at Week 4. 95% confidence interval estimate and p-value (based upon a normal approximation) were also computed from the LS mean differences and variability estimates from the model; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Difference in LS Means = 4.1, 95% CI 2-sided [1.3 to 6.9], Standard Error of Mean 1.42
Statistical Analysis 7: Comparison: Placebo vs MK-6096 10 mg; MK-6096 10 mg vs. Placebo at Week 4 A mixed effects model with terms for baseline value, geographic region (Japan vs. ex-Japan), gender, treatment, sequence, period, time, and treatment-by-time interaction and period-by-time interaction was used to estimate LS mean differences between MK-6096 and placebo at Week 4. 95% confidence interval estimate and p-value (based upon a normal approximation) were also computed from the LS mean differences and variability estimates from the model; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = 9.7, 95% CI 2-sided [6.9 to 12.5], Standard Error of Mean 1.43
Statistical Analysis 8: Comparison: Placebo vs MK-6096 20 mg; MK-6096 20 mg vs. Placebo at Week 4 A mixed effects model with terms for baseline value, geographic region (Japan vs. ex-Japan), gender, treatment, sequence, period, time, and treatment-by-time interaction and period-by-time interaction was used to estimate LS mean differences between MK-6096 and placebo at Week 4. 95% confidence interval estimate and p-value (based upon a normal approximation) were also computed from the LS mean differences and variability estimates from the model; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = 8.7, 95% CI 2-sided [5.9 to 11.5], Standard Error of Mean 1.43

2. Secondary Outcome: Wake After Persistent Sleep Onset (WASO) on Night 1 and After 4 Weeks of Treatment
Description: WASO was measured using a PSG, which consisted of an EEG for registration of brain activity during sleep, an EOG for registration of the eye movements during sleep, and an EMG for recording chin muscle activity during sleep. Sleep stage scoring was performed visually in 30-second epochs according to R&K criteria and PSG data were read by a Central Reader. WASO was defined as the duration of wakefulness measured in minutes (any epoch of Stage 0) from persistent sleep onset (first epoch of the first twenty consecutive epochs of non-wake) to lights on. LS mean WASO was reported for each treatment arm.
Time Frame: Night 1 and end of Week 4
Population: FAS population; subset of all randomized participants who received at least one dose of study medication and had any post-randomization WASO efficacy assessment data. The FAS population may have varied across endpoints due to the degree of missing data for each endpoint.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | MK-6096 2.5 mg | MK-6096 5 mg | MK-6096 10 mg | MK-6096 20 mg
Number analyzed (Participants) | 313 | 79 | 78 | 80 | 80
minutes
  Night 1 (n=313, 79, 78, 80, 80) | 83.1 (2.81) | 52.3 (6.11) | 50.6 (6.14) | 52.2 (6.06) | 37.3 (6.07)
  Week 4 (n=300, 76, 76, 76, 75) | 76.1 (2.77) | 60.6 (5.62) | 62.9 (5.62) | 50.5 (5.63) | 46.1 (5.65)
Statistical Analysis 1: Comparison: Placebo vs MK-6096 2.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = -30.8, 95% CI 2-sided [-43.2 to -18.4], Standard Error of Mean 6.29
Statistical Analysis 2: Comparison: Placebo vs MK-6096 5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = -32.5, 95% CI 2-sided [-44.9 to -20.1], Standard Error of Mean 6.31
Statistical Analysis 3: Comparison: Placebo vs MK-6096 10 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = -30.9, 95% CI 2-sided [-43.2 to -18.7], Standard Error of Mean 6.21
Statistical Analysis 4: Comparison: Placebo vs MK-6096 20 mg; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = -45.8, 95% CI 2-sided [-58.0 to -33.5], Standard Error of Mean 6.22
Statistical Analysis 5: Comparison: Placebo vs MK-6096 2.5 mg; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; Difference in LS Means = -15.5, 95% CI 2-sided [-26.7 to -4.4], Standard Error of Mean 5.65
Statistical Analysis 6: Comparison: Placebo vs MK-6096 5 mg; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; p = 0.020, Mixed Models Analysis; Difference in LS Means = -13.2, 95% CI 2-sided [-24.4 to -2.1], Standard Error of Mean 5.66
Statistical Analysis 7: Comparison: Placebo vs MK-6096 10 mg; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = -25.7, 95% CI 2-sided [-36.8 to -14.5], Standard Error of Mean 5.67
Statistical Analysis 8: Comparison: Placebo vs MK-6096 20 mg; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = -30.0, 95% CI 2-sided [-41.2 to -18.8], Standard Error of Mean 5.69

3. Secondary Outcome: Latency to the Onset of Persistent Sleep (LPS) on Night 1 and After 4 Weeks of Treatment
Description: LPS was measured using a PSG, which consisted of an EEG for registration of brain activity during sleep, an EOG for registration of the eye movements during sleep, and an EMG for recording chin muscle activity during sleep. Sleep stage scoring was performed visually in 30-second epochs according to R&K criteria and PSG data were read by a Central Reader. LPS was defined as the duration of time measured in minutes from lights off to persistent sleep onset. An epoch of non-wake was defined as a 30-second interval classified as either Stage 1, 2, 3, 4 or REM according to conventional R&K scoring. LS mean LPS was reported for each treatment arm.
Time Frame: Night 1 and end of Week 4
Population: FAS population; subset of all randomized participants who received at least one dose of study medication and had any post-randomization LPS efficacy assessment data. The FAS population may have varied across endpoints due to the degree of missing data for each endpoint.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | MK-6096 2.5 mg | MK-6096 5 mg | MK-6096 10 mg | MK-6096 20 mg
Number analyzed (Participants) | 313 | 79 | 78 | 80 | 80
minutes
  Night 1 (n=313, 79, 78, 80, 80) | 43.4 (2.06) | 33.2 (4.35) | 27.7 (4.36) | 19.9 (4.32) | 23.0 (4.31)
  Week 4 (n=300, 76, 76, 76, 75) | 39.4 (2.19) | 30.5 (4.55) | 30.7 (4.55) | 19.9 (4.57) | 28.1 (4.58)
Statistical Analysis 1: Comparison: Placebo vs MK-6096 2.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.022, Mixed Models Analysis; Difference in LS Means = -10.2, 95% CI 2-sided [-18.9 to -1.5], Standard Error of Mean 4.43
Statistical Analysis 2: Comparison: Placebo vs MK-6096 5 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = -15.7, 95% CI 2-sided [-24.5 to -7.0], Standard Error of Mean 4.44
Statistical Analysis 3: Comparison: Placebo vs MK-6096 10 mg; [analysis description as in outcome 1, analysis 3]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = -23.5, 95% CI 2-sided [-32.1 to -14.9], Standard Error of Mean 4.38
Statistical Analysis 4: Comparison: Placebo vs MK-6096 20 mg; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = -20.3, 95% CI 2-sided [-29.0 to -11.7], Standard Error of Mean 4.38
Statistical Analysis 5: Comparison: Placebo vs MK-6096 2.5 mg; [analysis description as in outcome 1, analysis 5]; Test type: Superiority or Other; p = 0.055, Mixed Models Analysis; Difference in LS Means = -8.9, 95% CI 2-sided [-18.0 to 0.2], Standard Error of Mean 4.61
Statistical Analysis 6: Comparison: Placebo vs MK-6096 5 mg; [analysis description as in outcome 1, analysis 6]; Test type: Superiority or Other; p = 0.060, Mixed Models Analysis; Difference in LS Means = -8.7, 95% CI 2-sided [-17.8 to 0.4], Standard Error of Mean 4.61
Statistical Analysis 7: Comparison: Placebo vs MK-6096 10 mg; [analysis description as in outcome 1, analysis 7]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Difference in LS Means = -19.5, 95% CI 2-sided [-28.6 to -10.4], Standard Error of Mean 4.62
Statistical Analysis 8: Comparison: Placebo vs MK-6096 20 mg; [analysis description as in outcome 1, analysis 8]; Test type: Superiority or Other; p = 0.015, Mixed Models Analysis; Difference in LS Means = -11.3, 95% CI 2-sided [-20.5 to -2.2], Standard Error of Mean 4.63

4. Primary Outcome: Percentage of Participants With at Least One Adverse Event (AE) During Treatment Periods 1 and 2
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product, was also an AE. The percentage of participants with AEs are presented for the first day of randomized treatment dosing (Day 1) through the last day of randomized treatment dosing (Day 29) in Treatment Periods 1 and 2.
Time Frame: Day 1 through Day 29 in Treatment Periods 1 and 2 (58 days total)
Population: All Participants as Treated (APaT) population; all randomized participants who received at least one dose of study treatment. Participants were included corresponding to the study treatment they actually received for a given period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | MK-6096 2.5 mg | MK-6096 5 mg | MK-6096 10 mg | MK-6096 20 mg
Number analyzed (Participants) | 315 | 79 | 78 | 80 | 81
percentage of participants | 26.0 | 26.6 | 25.6 | 32.5 | 34.6
Statistical Analysis 1: Comparison: Placebo vs MK-6096 2.5 mg; Miettinen and Nurminen's method was used to calculate confidence intervals for between-treatment differences in the percentage of participants with events versus placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-9.5 to 12.2]
Statistical Analysis 2: Comparison: Placebo vs MK-6096 5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-10.3 to 11.2]
Statistical Analysis 3: Comparison: Placebo vs MK-6096 10 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 6.5, 95% CI 2-sided [-4.2 to 18.3]
Statistical Analysis 4: Comparison: Placebo vs MK-6096 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 8.5, 95% CI 2-sided [-2.3 to 20.4]

5. Primary Outcome: Percentage of Participants That Discontinued Study Medication Due to an AE During Treatment Periods 1 and 2
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which is temporally associated with the use of the SPONSOR's product, was also an AE. The percentage of participants that discontinued study medication due to AEs are presented for the first day of randomized treatment dosing (Day 1) through the last day of randomized treatment dosing (Day 29) in Treatment Periods 1 and 2.
Time Frame: Day 1 through Day 29 in Treatment Periods 1 and 2 (58 days total)
Population: APaT population; all randomized participants who received at least one dose of study treatment. Participants were included corresponding to the study treatment they actually received for a given period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | MK-6096 2.5 mg | MK-6096 5 mg | MK-6096 10 mg | MK-6096 20 mg
Number analyzed (Participants) | 315 | 79 | 78 | 80 | 81
percentage of participants | 2.2 | 5.1 | 1.3 | 2.5 | 0.0
Statistical Analysis 1: Comparison: Placebo vs MK-6096 2.5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-1.0 to 10.2]
Statistical Analysis 2: Comparison: Placebo vs MK-6096 5 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-3.6 to 4.8]
Statistical Analysis 3: Comparison: Placebo vs MK-6096 10 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-2.7 to 6.6]
Statistical Analysis 4: Comparison: Placebo vs MK-6096 20 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-4.5 to 2.3]

ADVERSE EVENTS:
Time Frame: From time of first dose through follow-up (up to 86 days)
Description: APaT population; all randomized participants who received ≥1 dose of study treatment. Participants in a treatment arm were counted once for each therapy received during a Treatment Period (TP), and the same participant may have been counted twice: once for the therapy assigned for TP 1 and once for the therapy assigned for TP2.
Groups:
- Washout: Participants administered single-blind placebo study medication for the first 3 nights of the washout period that occurred between Treatment Period 1 and Treatment Period 2, immediately prior to bedtime. The remaining 11 days of the washout period constituted a drug holiday during which time no study medication was administered.
- Post-Study/Follow-up: Participants that completed the study or prematurely discontinued during either treatment period received a 14-day (from last dose) follow-up phone call to assess for AEs. The Post-Study/Follow-up period was the period that occurred between study completion/ treatment discontinuation and the 14-day follow-up phone call (14 days after the last dose of double-blind study medication).
Arm/Group | Placebo | MK-6096 2.5 mg | MK-6096 5 mg | MK-6096 10 mg | MK-6096 20 mg | Washout | Post-Study/Follow-up
Serious Adverse Events (participants affected / at risk) | 0/315 | 1/79 | 1/78 | 1/80 | 0/81 | 1/315 | 1/324
Other Adverse Events (participants affected / at risk) | 21/315 | 3/79 | 5/78 | 10/80 | 14/81 | 5/315 | 0/324
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=315) | MK-6096 2.5 mg (N=79) | MK-6096 5 mg (N=78) | MK-6096 10 mg (N=80) | MK-6096 20 mg (N=81) | Washout (N=315) | Post-Study/Follow-up (N=324)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=315) | MK-6096 2.5 mg (N=79) | MK-6096 5 mg (N=78) | MK-6096 10 mg (N=80) | MK-6096 20 mg (N=81) | Washout (N=315) | Post-Study/Follow-up (N=324)
Headache (Nervous system disorders) | 12 (14) | 3 (3) | 3 (4) | 5 (5) | 3 (3) | 4 (4) | 0 (0)
Somnolence (Nervous system disorders) | 9 (9) | 1 (1) | 2 (2) | 5 (6) | 11 (13) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less